CLINICAL TRIAL: NCT02324946
Title: Comparison of STOP-BANG and DES-OSA as Predictive Score for Difficult Intubation Among Patients Scheduled for Bariatric Surgery.
Brief Title: Comparison of STOP-BANG and DES-OSA as Predictive Score for Difficult Intubation.
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Eric Deflandre, MD, FCCP, Astes
Other Study IDs: STOP-BANG, DES-OSA
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Bariatric Surgery Candidate
Keywords: Sleep Apnea Syndromes; Perioperative Period; Mass Screening
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Mass Screening
  Interventions: Other: Mass Screening

INTERVENTIONS:
Other: Mass Screening — Preoperative screening with STOP-BANG and DES-OSA scores and postoperative comparison with difficult intubation / ventilation scores.

SUMMARY:
The DES-OSA Score and the STOP-BANG score were predictive scores for Obstructive Sleep Apnea.

This study will compare, among patients scheduled for bariatric surgery, these two scores as predictive scores for a difficult intubation.

DETAILED DESCRIPTION:
The DES-OSA Score and the STOP-BANG score were predictive scores for Obstructive Sleep Apnea.

This study will compare, among patients scheduled for bariatric surgery, these two scores as predictive scores for a difficult mask ventilation of tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg m-2
* Preoperative Polysomnography

Exclusion Criteria:

* Pregnant women
* ENT Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for bariatric surgery
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Predictive value of STOP-BANG and DES-OSA scores for difficult mask ventilation or intubation. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Eric P DEFLANDRE, MD, FCCP, Study Chair — Astes
Locations (1):
- Clinique Saint-Luc de Bouge, Bouge, Namur, Belgium